CLINICAL TRIAL: NCT02606773
Title: Open-label, Randomized Comparator Study for Evaluation the Bioavailability of "Novo C Plus" Vitamin C Containing Dietary Supplement in Healthy Subjects
Brief Title: "Novo C Plus" Vitamin C Containing Dietary Supplement Bioavailability in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Novonex Pharma Kft (Industry)
Responsible Party: Principal Investigator, Istvan Takacs, Reader in university, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVP-14C
Record Dates: First submitted 2015-11-13; First posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Vitamin C Deficiency
Keywords: vitamin C supplementation
MeSH Terms: conditions — Ascorbic Acid Deficiency | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 600 mg Novo C plus (Experimental): Single dose of oral 600 mg Novo C plus dietary supplement (contains 600 mg ascorbic acid in liposomal formulation)
  Interventions: Drug: Ascorbic Acid
- 900 mg Novo C Plus (Experimental): Single dose of 900 mg oral Novo C plus dietary supplement (contains 900 mg ascorbic acid in liposomal formulation)
  Interventions: Drug: Ascorbic Acid
- 500 mg intravenous vitamin C (Active Comparator): Single dose of 500 mg intravenous ascorbic acid (Vitamin C 100 mg/ml injection; EGIS)
  Interventions: Drug: Ascorbic Acid
- 500 mg oral vitamin C (Active Comparator): Single dose of 500 mg oral ascorbic acid (Cetebe 500 mg retard capsules; GlaxoSmithKline Consumer Healthcare - GSK Export)
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — Ascorbic acid in different ways and doses

SUMMARY:
The aim of this study is to evaluate the bioavailability of "Novo C Plus" vitamin C containing dietary supplement compared to licensed vitamin C medications. The novelty of this product is the liposomal formulation.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years old healthy volunteers
* body weight >45 kg
* body height >150 cm
* plasma ascorbic acid at screening <75 µmol/l
* signed written informed consent
* subject agrees avoid vitamin C containing medications and dietary supplements from screening until V0 visit (maximum 15 days)
* subject agrees to avoid high activity physical exercise 72 hours prior to V0 visit

Exclusion Criteria:

* confirmed or suspected active infection
* liver or renal failure (equal or greater than CKD3)
* chronic disease that affects absorption or vitamin C metabolism
* severe metabolic disorder
* body mass index >35 kg/m2
* malabsorption syndrome that affects vitamin C metabolism
* heart failure, angina pectoris, ventricular arrhythmias or atrial fibrillation with >100/min ventricular rate
* gastrointestinal bleeding in past three months
* uncontrolled diabetes mellitus (HbA1c>8,5%)
* malignant disease
* alcohol or drug abuse
* active psychiatric disorder, intention for suicidal, disorders with unconsciousness
* psychopathic disorder, lack of cooperation
* known coagulopathy
* chronic obstructive lung disease or active smoking (more than 2 cigarettes in the past 6 months)
* untreated hypertension if blood pressure is greater than 165/95 mmHg
* gravidity or breastfeeding
* taking more than 100 mg vitamin C daily within 2 weeks to screening

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Plasma ascorbic acid concentration area under curve | 360 minutes
  Plasma ascorbic acid concentration will be measured from peripheral blood samples after 30-45-60-90-120-180-240-300-360 minutes after getting the medication. Area under curve of time - plasma concentration curve will be calculated.

SECONDARY OUTCOMES:
Safety and tolerability assessed by number of subjects with treatment-related adverse events as assessed by CTCAE v4.0 | 24 hours
Urine ascorbic acid excretion | 12 hours
  Urine is collected for 12 hours after taking study drug, and urine ascorbic acid excretion will be calculated: urine ascorbic acod concentration (uM)×collected urine (L).

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University - 1st Departement of Internal Medicine, Budapest, Hungary